CLINICAL TRIAL: NCT02007512
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY OF EFFICACY AND SAFETY OF ENZALUTAMIDE IN COMBINATION WITH EXEMESTANE IN PATIENTS WITH ADVANCED BREAST CANCER THAT IS ESTROGEN OR PROGESTERONE RECEPTOR-POSITIVE AND HER2-NORMAL
Brief Title: Efficacy and Safety Study of Enzalutamide in Combination With Exemestane in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDV3100-12; 2013-002717-35 (EudraCT Number); C3431008 (Other: Alias Study Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-10 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: advanced breast cancer; enzalutamide; MDV3100; Estrogen receptor positive (ER +); Progesterone receptor positive (PgR +); HER-2 normal
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzalutamide & exemestane (Experimental): Enzalutamide 160 mg/day administered as four 40mg soft gelatin capsules by mouth once daily with or without food and exemestane 50mg (two 25mg tablets overencapsulated as a single capsule during the blinded portion of the study and two 25mg tablets after unblinding) once daily after food.
  Interventions: Drug: Enzalutamide; Drug: exemestane
- Placebo & exemestane (Active Comparator): Placebo and exemestane 25mg (overencapsulated to match 50mg dose during the blinded portion of the study and one 25mg tablet without placebo after unblinding) once daily after food.
  Interventions: Drug: exemestane; Drug: Placebo (for enzalutamide)

INTERVENTIONS:
Drug: Enzalutamide — 160 mg/day administered as four 40mg soft gelatin capsules by mouth once daily with or without food.
  Other Names: MDV3100; XTANDI
  Arms: Enzalutamide & exemestane
Drug: exemestane — 25mg (overencapsulated to match 50mg dose during the blinded portion of the study and one 25mg tablet after unblinding) by mouth once daily after food.
  Other Names: Aromasin
  Arms: Placebo & exemestane
Drug: Placebo (for enzalutamide) — Sugar pill manufactured to mimic enzalutamide administered as four soft gelatin capsules by mouth once daily with or without food.
  Arms: Placebo & exemestane
Drug: exemestane — 50mg (two 25mg tablets overencapsulated as a single capsule during the blinded portion of the study and two 25mg tablets after unblinding) by mouth once daily after food.
  Other Names: Aromasin
  Arms: Enzalutamide & exemestane

SUMMARY:
The purpose of this study is to determine if enzalutamide given in combination with exemestane is safe and effective in patients with advanced breast cancer.

DETAILED DESCRIPTION:
This is a Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Efficacy and Safety of Enzalutamide in Combination With Exemestane in Patients With Advanced Breast Cancer That Is Estrogen or Progesterone Receptor Positive and HER2-Normal.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Postmenopausal;
* Advanced histologically confirmed breast cancer that is ER+, PgR+, or both, and HER-2 normal;
* Up to one prior hormone therapy and up to one prior chemotherapy in the advanced setting is allowed;
* Availability of a representative, formalin-fixed, paraffin-embedded tumor specimen that enabled the diagnosis of breast cancer with viable tumor cells in a tissue block or unstained serial slides accompanied bay an associated pathology report;
* Measurable disease. Patients with non-measurable bone or skin disease as their only manifestation of advanced breast cancer are also eligible;
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1;

Exclusion Criteria:

* Any severe concurrent disease, infection, or comorbid condition that renders the patient inappropriate for enrollment in the opinion of the investigator;
* Any condition or reason that interferes with the patient's ability to participate in the trial, that may cause undue risk, or complicates the interpretation of safety data, in the opinion of the investigator;
* Current or previously treated brain metastasis or leptomeningeal disease;
* Prior therapy (> 28 days) with exemestane in the metastatic setting (Patients receiving exemestane in the adjuvant setting and having disease recurrence more than 1 year after treatment discontinuation are eligible);
* Requires treatment for tuberculosis or HIV infection;
* Radiation therapy within 7 days before randomization;
* History of another invasive cancer within 5 years before randomization;
* History of seizure or any condition that may predispose to seizure;
* Clinically significant cardiovascular disease;
* Active gastrointestinal disorder;
* Major surgery within 28 days prior to randomization;
* Treatment with any oral anticancer or with any non-hormonal anticancer agent within 14 days before randomization;
* Treatment with any approved or investigational agent that blocks androgen synthesis or targets the androgen receptor;
* Treatments with any of the following medications within 14 days before randomization: Estrogens, Androgens, or Systemic radionuclides;
* Hypersensitivity reaction to exemestane.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 247 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (115):
- United States (78):
  - ATTN-Research Pharmacist, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Anschutz Outpatient Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Englewood, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists, Hudson, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center,, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Clinic, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology Hematology, P.A, Minneapolis, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health System DBA Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Dr.Michaela Tsai, Minneapolis, Minnesota
  - The West Clinic, P.C., Corinth, Mississippi
  - The West Clinic, P.C. d/b/a West Cancer Center, Southaven, Mississippi
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center- West County, St Louis, Missouri
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oncology Hematology Care, Inc., Fairfield, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Greenville Health System, Seneca, South Carolina
  - Greenville Health System, Spartanburg, South Carolina
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - The West Clinic, P.C. d/b/a West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - The West Clinic, P.C. d/b/a West Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt Health Pharmacy One Hundred Oaks, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Institute, Mechanicsville, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
- Belgium (3):
  - UZA, Edegem, Antwerpen
  - GZA, Wilrijk, Antwerpen
  - Institut Jules Bordet, Brussels
- Canada (3):
  - Sunnybrook Research Institute, Toronto, Ontario
  - McGill University Health Center- Cedars Cancer Center, Montreal, Quebec
  - McGill University Health Centre - Cedars Cancer Centre, Montreal, Quebec
- Ireland (6):
  - Pharmacy Department, Dublin
  - Radiology Department, Dublin
  - St Vincent's University Hospital, Dublin
  - Institute for Cancer Research, Dublin
  - Mater Private Hospital, Dublin
  - Cancer Clinical Trials Unit, Dublin
- Italy (7):
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Divisione di Senologia Medica; Istituto Europeo di Oncologia, Milan, MI
  - A.O.di Perugia S. Maria Della Misericoridia, Perugia, PG
  - Azienda Ospedaliera S.Orsola Malpighi, Bologna
  - U.O. Farmaceutica, Nuovo Ospedale di Prato, Prato
  - U.O. Oncologia Medica, Nuovo Ospedale di Prato, Prato
  - Dipartimento di Oncologia Medica, Istituto Nazionale Tumori Regina Elena, Roma
- Spain (7):
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Grupo Hospitalario Quiron - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital de Madrid Norte Sanchinarro, Madrid
- United Kingdom (11):
  - Brighton and Sussex University Hospital NHS Trust, Brighton, England
  - Pharmacy Department, Brighton, England
  - Radiation Safety Service, Medical Physics Department, Brighton, England
  - Histopathology Department, Nottingham, England
  - Nottingham University Hospital, Nottingham, England
  - Pharmacy Department, Nottingham, England
  - Radiology Department, Nottingham, England
  - Department of Radiology, Truro, England
  - Pharmacy Department, Truro, England
  - Royal Cornwall Hospitals NHS trust, Truro, England
  - Clinical Investigation & Research Unit, Brighton, Sussex

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 247 participants were enrolled.
Pre-assignment Details: This was a phase 2, randomized, double blind, placebo-controlled study.
Groups:
- Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg: Participants with no previous hormonal treatment for advanced breast cancer, received enzalutamide 160 mg along with exemestane 50 mg, orally, once daily until disease progression or permanent treatment discontinuation. Participants were followed-up until 30 days after last dose of study drug, death, or before initiation of a new antitumor treatment, whichever occurred first.
- Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg: Participants with previous disease progression following hormonal treatment for advanced breast cancer, received enzalutamide 160 mg along with exemestane 50 mg, orally, once daily in double blind treatment period until disease progression or permanent treatment discontinuation. Participants were followed-up until 30 days after last dose of study drug, death, or before initiation of a new antitumor treatment, whichever occurred first.
- Cohort 1: Placebo + Exemestane 25 mg: Participants with no previous hormonal treatment for advanced breast cancer received placebo matched to enzalutamide along with exemestane 25 mg, orally, once daily in double blind treatment period until disease progression or permanent treatment discontinuation. Eligible participants with disease progression in double blind period, on their discretion, received enzalutamide 160 mg along with exemestane 50 mg, orally, once daily up to disease progression in open label treatment period. Participants were followed-up until 30 days after last dose of study drug, death, or before initiation of a new antitumor treatment, whichever occurred first.
- Cohort 2: Placebo + Exemestane 25 mg: Participants with previous disease progression following hormonal treatment for advanced breast cancer, received placebo matched to enzalutamide along with exemestane 25 mg, orally, once daily in double blind treatment period until disease progression or permanent treatment discontinuation. Eligible participants with disease progression in double blind period, on their discretion, received enzalutamide 160 mg along with exemestane 50 mg, orally, once daily up to disease progression in open label treatment period. Participants were followed-up until 30 days after last dose of study drug, death, or before initiation of a new antitumor treatment, whichever occurred first.
Period: Double Blind Treatment Period
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Placebo + Exemestane 25 mg
Started | 63 | 60 | 64 | 60
Treated | 62 | 60 | 63 | 60
Completed | 0 | 0 | 0 | 0
Not Completed | 63 | 60 | 64 | 60
Not completed — Adverse Event | 4 | 6 | 2 | 2
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Disease progression | 51 | 50 | 57 | 52
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Other | 2 | 1 | 1 | 2
Not completed — Randomized but not treated | 1 | 0 | 1 | 0
Period: Open Label Treatment Period
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Placebo + Exemestane 25 mg
Started | 25 | 12 | 0 | 0
Treated | 24 | 11 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 25 | 12 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0
Not completed — Disease progression | 23 | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the participants randomly assigned to double-blind study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg | Total
Number analyzed (Participants) | 63 | 64 | 60 | 60 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 32 | 37 | 40 | 151
  >=65 years | 21 | 32 | 23 | 20 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 64 | 60 | 60 | 247
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS): Intent-to-Treat (ITT) Population By Interactive Web Recognition System (IWRS)
Description: PFS was defined as the time in months from randomization to the first documentation of progression of disease (PD) or death on study due to any cause, whichever occurred first. PD according to response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) was defined as greater than or equal to (>=) 20 percent (%) increase in the sum of diameters of the target lesions taking as a reference the smallest sum recorded since the start of treatment or unequivocal progression in non-target lesions or the appearance of 1 or more new lesions. The analysis of PFS was based on investigator assessment of disease progression. Participants who were not known to have had a PFS event at the analysis date were censored at last tumor assessment date prior to data cutoff or date of new treatment initiation, whichever occurred first.
Time Frame: From randomization until PD, last tumor assessment without PD before new antitumor treatment initiation or death due to any cause, whichever occurred first (up to 3 years)
Population: ITT population included all the participants randomly assigned to double-blind study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 63 | 64 | 60 | 60
months | 11.8 [7.3 to 15.9] | 5.8 [3.5 to 10.9] | 3.6 [1.9 to 5.5] | 3.9 [2.6 to 5.4]
Statistical Analysis 1: Comparison: Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 1: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.3631, Stratified log-rank; Hazard Ratio (HR) = 0.820, 95% CI 2-sided [0.535 to 1.257]
Statistical Analysis 2: Comparison: Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 2: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.9212, Stratified log-rank; Hazard Ratio (HR) = 1.022, 95% CI 2-sided [0.659 to 1.586]

2. Primary Outcome: Progression Free Survival (PFS): Diagnostic Positive (DX+) Population By Interactive Web Recognition System (IWRS)
Description: PFS was defined as the time in months from randomization to the first documentation of PD or death on study due to any cause, whichever occurred first. PD according to RECIST 1.1, was defined as >= 20% increase in the sum of diameters of the target lesions taking as a reference the smallest sum recorded since the start of treatment or unequivocal progression in non-target lesions or the appearance of 1 or more new lesions. The analysis of PFS was based on investigator assessment of disease progression. Participants who were not known to have had a PFS event at the analysis date were censored at last tumor assessment date prior to data cutoff or date of new treatment initiation, whichever occurred first.
Time Frame: as for outcome 1
Population: Dx+ population: Subset of ITT population, defined prior to the first unblinded analysis as meeting the threshold for diagnostic score based on ribonucleic acid (RNA) sequencing data from tumor tissue. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 24 | 26 | 15 | 20
months | 16.5 [11.0 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016). | 4.3 [1.9 to 10.9] | 6.0 [2.3 to 26.7] | 5.3 [1.8 to 6.7]
Statistical Analysis 1: Comparison: Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 1: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.0335, Stratified log-rank; Hazard Ratio (HR) = 0.442, 95% CI 2-sided [0.205 to 0.955]
Statistical Analysis 2: Comparison: Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 2: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.1936, Stratified log-rank; Hazard Ratio (HR) = 0.554, 95% CI 2-sided [0.225 to 1.363]

3. Secondary Outcome: Clinical Benefit Rate-24 (CBR-24)
Description: CBR-24: Percentage of participants with a best response of complete response (CR), partial response (PR), or stable disease (SD) sustained for atleast 24 weeks, as determined by investigator using RECIST 1.1. CR: Disappearance of all (target and non-target) lesions and normalization of tumor marker level for non-target lesions. All lymph nodes (target and non-target) must be non-pathological in size (less than [<] 10 millimeter [mm] short axis). PR: >=30% decrease in sum of diameters of target lesions, using baseline sum diameters as reference. SD: Neither sufficient reduction to qualify as PR nor sufficient increase to qualify as PD, using the smallest sum diameters during study as reference. PD: >=20% increase (an absolute increase of >=5 mm) in sum of diameters of target lesions, using the smallest sum during the study as a reference (including baseline sum), or unequivocal progression of existing non-target lesions, or appearance of atleast 1 new target or non-target lesions.
Time Frame: From randomization up to 3 years
Population: ITT population included all the participants randomly assigned to double-blind study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 63 | 64 | 60 | 60
percentage of participants | 61.9 [48.8 to 73.9] | 45.3 [32.8 to 58.3] | 20.0 [10.8 to 32.3] | 31.7 [20.3 to 45.0]

4. Secondary Outcome: Best Objective Response Rate
Description: Best objective response rate: Percentage of participants with measurable disease and with a best response of CR or PR according to RECIST 1.1. CR: Disappearance of all (target and non-target) lesions and normalization of tumor marker level for non-target lesions. All lymph nodes (target and non-target) must be non-pathological in size (<10 mm short axis). PR: Atleast 30% decrease in sum of diameters of target lesions, using baseline sum diameters as reference. Response evaluation was based on investigators' judgment.
Time Frame: From randomization until CR or PR, whichever occurred first (up to 3 years)
Population: ITT population included all the participants randomly assigned to double-blind study treatment. Here 'Number of participants analyzed' signifies participants with measurable response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 39 | 42 | 42 | 42
percentage of participants | 30.8 [17.0 to 47.6] | 19.0 [8.6 to 34.1] | 9.5 [2.7 to 22.6] | 4.8 [0.6 to 16.2]

5. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response: Time from first documentation of CR or PR, to the first documentation of PD or death due to any cause, whichever occurred first as determined by investigator using RECIST 1.1. CR: Disappearance of all (target and non-target) lesions and normalization of tumor marker level for non-target lesions. All lymph nodes (target and non-target) must be non-pathological in size (<10 mm short axis). PR: >=30% decrease in sum of diameters of target lesions, using baseline sum diameters as reference. PD: >=20% increase (an absolute increase of >=5 mm) in sum of diameters of target lesions, using the smallest sum during the study as a reference (including baseline sum), or unequivocal progression of existing non-target lesions, or appearance of atleast 1 new target or non-target lesions. Participants with no PD or death (after initial CR or PR) at the analysis date were censored at last tumor assessment date prior to date of new antitumor treatment or data cutoff.
Time Frame: From first documentation of CR or PR until PD, or last tumor assessment without PD before new antitumor treatment initiation or death due to any cause, whichever occurred first (up to 3 years)
Population: ITT population included all the participants randomly assigned to double-blind study treatment. Here 'Number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 39 | 42 | 42 | 42
months | 14.0 [5.6 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016). | 9.1 [3.2 to 10.2] | 18.3 [3.3 to 23.1] | 4.6 [1.9 to 7.4]

6. Secondary Outcome: Time to Response
Description: Time to response: Time from randomization to first documentation of CR or PR. CR: Disappearance of all (target and non-target) lesions and normalization of tumor marker level for non-target lesions. All lymph nodes (target and non-target) must be non-pathological in size (<10 mm short axis). PR: >=30% decrease in sum of diameters of target lesions, using baseline sum diameters as reference. PD: >=20% increase (an absolute increase of >=5 mm) in sum of diameters of target lesions, using the smallest sum during the study as a reference (including baseline sum), or unequivocal progression of existing non-target lesions, or appearance of atleast 1 new target or non-target lesions. Participants who were not known to have had a CR or PR were censored at last tumor assessment date prior to data cutoff or date of new treatment initiation, whichever occurred first.
Time Frame: From randomization until first documentation of CR or PR, or last tumor assessment without PD or death prior to new antitumor treatment initiation, whichever occurred first (up to 3 years)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 39 | 42 | 42 | 42
months | 12.9 [7.3 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016). | 14.0 [7.4 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016). | NA [3.9 to NA] — Median and upper limit of 95% confidence interval were not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016). | NA [NA to NA] — Median and 95% confidence interval were not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016).

7. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from the date of randomization to PD defined by the investigator using RECIST 1.1. PD: >=20% increase (an absolute increase of >=5 mm) in sum of diameters of target lesions, using the smallest sum during the study as a reference (including baseline sum), or unequivocal progression of existing non-target lesions, or appearance of atleast 1 new target or non-target lesions. Participants who did not experience disease progression, time to progression was right censored at the date of the last tumor assessment prior to data cutoff or date of new antitumor treatment, whichever occurred first.
Time Frame: From randomization until PD or last tumor assessment without PD before new antitumor treatment initiation, whichever occurred first (up to 3 years)
Population: ITT population included all the participants randomly assigned to double-blind study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 63 | 64 | 60 | 60
months | 11.8 [7.3 to 15.9] | 7.4 [3.5 to 13.5] | 3.6 [1.9 to 5.6] | 3.9 [2.6 to 5.4]

8. Secondary Outcome: Progression Free Survival (PFS) at 6 Months
Description: PFS at 6 months was defined as the percentage of participants with no event of disease progression at Month 6 landmark, estimated by Kaplan-Meier methods. PFS was defined as the time in months from randomization to the first documentation of PD or death on study due to any cause, whichever occurred first. PD: >=20% increase (an absolute increase of >=5 mm) in sum of diameters of target lesions, using the smallest sum during the study as a reference (including baseline sum), or unequivocal progression of existing non-target lesions, or appearance of atleast 1 new target or non-target lesions. The analysis of PFS was based on investigator assessment of disease progression.
Time Frame: Month 6
Population: ITT population included all the participants randomly assigned to double-blind study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 63 | 64 | 60 | 60
percentage of participants | 66.7 [53.2 to 77.0] | 50.0 [37.1 to 61.6] | 31.5 [19.7 to 43.9] | 33.3 [21.6 to 45.5]

9. Secondary Outcome: Concentration Versus Time Summary of Enzalutamide
Description: Concentration versus time summary was calculated by setting concentration values below limit of quantitation to zero.
Time Frame: Predose on Day 29, 57 and 113
Population: Pharmacokinetic (PK) population for enzalutamide included all participants in safety population who received any amount of enzalutamide and had at least 1 reportable concentration value for enzalutamide or its active metabolite (N-desmethyl enzalutamide).
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Groups:
- Enzalutamide 160 mg: Participants received enzalutamide 160 mg dose orally, once daily, either in double blind treatment period or in open label treatment period until disease progression or permanent treatment discontinuation. Participants were followed-up until 30 days after the last dose of study drug, death, or before initiation of a new antitumor treatment, whichever occurred first.
Arm/Group | Enzalutamide 160 mg
Number analyzed (Participants) | 114
microgram per milliliter
  Day 29: number analyzed (Participants) | 109
  Day 29 | 14.2 (2.97)
  Day 57: number analyzed (Participants) | 92
  Day 57 | 14.2 (3.21)
  Day 113: number analyzed (Participants) | 67
  Day 113 | 13.2 (4.51)

10. Secondary Outcome: Concentration Versus Time Summary of Exemestane
Description: Concentration versus time summary was calculated by setting concentration values below limit of quantitation to zero.
Time Frame: Predose, 1 and 6 hour postdose on Day 29, 57, 113 and 169
Population: PK population for exemestane was defined as all participants in the safety population who received any amount of exemestane and had at least 1 reportable plasma concentration value for exemestane.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Groups:
- Exemestane 25 mg: Participants received exemestane 25 mg dose orally, once daily in double blind treatment period until disease progression or permanent treatment discontinuation. Participants were followed-up until 30 days after the last dose of study drug, death, or before initiation of a new antitumor treatment, whichever occurred first.
- Exemestane 50 mg: Participants received exemestane 50 mg dose orally, once daily until disease progression or permanent treatment discontinuation, either in double blind treatment period or in open label treatment period. Participants were followed-up until 30 days after the last dose of study drug, the date of death, or before initiation of a new antitumor treatment, whichever occurred first.
Arm/Group | Exemestane 25 mg | Exemestane 50 mg
Number analyzed (Participants) | 114 | 115
Picogram per milliliter
  Day 29: Predose: number analyzed (Participants) | 108 | 108
  Day 29: Predose | 1010 (1600) | 943 (939)
  Day 29: 1 hour Postdose: number analyzed (Participants) | 99 | 102
  Day 29: 1 hour Postdose | 17000 (16400) | 19200 (17800)
  Day 29: 6 hour Postdose: number analyzed (Participants) | 57 | 55
  Day 29: 6 hour Postdose | 5590 (4750) | 6850 (9090)
  Day 57: Predose: number analyzed (Participants) | 89 | 92
  Day 57: Predose | 1160 (2590) | 1100 (2650)
  Day 57: 1 hour Postdose: number analyzed (Participants) | 76 | 83
  Day 57: 1 hour Postdose | 19900 (18600) | 15300 (14500)
  Day 57: 6 hour Postdose: number analyzed (Participants) | 26 | 23
  Day 57: 6 hour Postdose | 5890 (4880) | 5650 (6200)
  Day 113: Predose: number analyzed (Participants) | 65 | 68
  Day 113: Predose | 1160 (2870) | 1330 (3380)
  Day 113: 1 hour Postdose: number analyzed (Participants) | 58 | 58
  Day 113: 1 hour Postdose | 20800 (18100) | 19400 (18500)
  Day 113: 6 hour Postdose: number analyzed (Participants) | 12 | 14
  Day 113: 6 hour Postdose | 3510 (3850) | 5600 (5290)
  Day 169: Predose: number analyzed (Participants) | 0 | 0
  Day 169: 1 hour Postdose: number analyzed (Participants) | 0 | 1
  Day 169: 1 hour Postdose |  | 22800 (NA) — Standard deviation could not be estimated since only 1 participant was analyzed.
  Day 169: 6 hour Postdose: number analyzed (Participants) | 0 | 1
  Day 169: 6 hour Postdose |  | 6020 (NA) — Standard deviation could not be estimated since only 1 participant was analyzed.

11. Secondary Outcome: Concentration Versus Time Summary of N-desmethyl Enzalutamide
Description: N-desmethyl enzalutamide was the active metabolite of enzalutamide. Concentration versus time summary was calculated by setting concentration values below limit of quantitation to zero.
Time Frame: Predose on Day 29, 57 and 113
Population: PK population for N-desmethyl enzalutamide included all the participants in safety population who received any amount of enzalutamide and had at least 1 reportable concentration value for N-desmethyl enzalutamide.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Enzalutamide 160 mg
Number analyzed (Participants) | 114
microgram per milliliter
  Day 29: number analyzed (Participants) | 109
  Day 29 | 11.6 (4.10)
  Day 57: number analyzed (Participants) | 92
  Day 57 | 15.2 (4.76)
  Day 113: number analyzed (Participants) | 67
  Day 113 | 15.2 (5.81)

12. Other Pre Specified Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Core Questionnaire (QLQ-C30) at Weeks 5, 9, 17, 25, 33, 41, 49, 61, 73, 85, 97, 109, 121 and 133: Global Health/Quality of Life
Description: The EORTC QLQ-C30 questionnaire was a standardized instrument developed to assess the quality of life of people with cancer. Participants self-rated their self-care, activity level, pain/discomfort, and mental health during the past week by choosing 1 of 4 possible responses that recorded the level of intensity (not at all, a little, quite a bit, and very much) within each dimension, where higher score=more level of intensity. The questionnaire also asked the participants to rate their overall health or quality of life within the past week on a scale of 1 to 7, where 1 is "very poor" and 7 is "excellent". Higher global health or quality of life scores indicated better overall health or quality of life. In this outcome measure, global health/quality of life scores are presented.
Time Frame: Baseline; Weeks 5, 9, 17, 25, 33, 41, 49, 61, 73, 85, 97, 109, 121 and 133
Population: ITT population included all the participants randomly assigned to double-blind study treatment. Here, "Overall Number of Participants Analyzed" contributed data to table but may not have evaluable data for every row and "Number Analyzed" signifies participants evaluable for the specified rows and value as "0" indicated no participants filled the questionnaire for the specified reporting group at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 63 | 60 | 60
Units on a scale
  Week 5: number analyzed (Participants) | 55 | 56 | 53 | 55
  Week 5 | 1.2 (19.14) | 1.3 (21.19) | -4.6 (16.55) | 0.3 (15.87)
  Week 9: number analyzed (Participants) | 54 | 50 | 43 | 44
  Week 9 | -1.9 (21.21) | 1.3 (18.77) | -5.6 (19.13) | -1.3 (14.37)
  Week 17: number analyzed (Participants) | 42 | 38 | 25 | 30
  Week 17 | -3.0 (19.46) | -1.8 (19.29) | -7.3 (24.45) | -0.8 (15.98)
  Week 25: number analyzed (Participants) | 37 | 34 | 15 | 21
  Week 25 | 3.6 (18.17) | -3.4 (21.03) | 0.6 (18.76) | -4.8 (16.79)
  Week 33: number analyzed (Participants) | 34 | 29 | 9 | 15
  Week 33 | 2.2 (19.60) | -0.9 (19.59) | -8.3 (17.68) | -5.0 (15.04)
  Week 41: number analyzed (Participants) | 29 | 22 | 9 | 12
  Week 41 | -0.9 (16.11) | -1.5 (16.99) | -9.3 (17.40) | -1.4 (9.95)
  Week 49: number analyzed (Participants) | 25 | 21 | 7 | 8
  Week 49 | -0.7 (19.53) | 0.8 (13.67) | -8.3 (12.73) | -4.2 (16.06)
  Week 61: number analyzed (Participants) | 22 | 19 | 7 | 4
  Week 61 | 3.8 (18.32) | -5.7 (19.26) | -1.2 (20.65) | 6.3 (18.48)
  Week 73: number analyzed (Participants) | 15 | 13 | 7 | 4
  Week 73 | -1.1 (19.64) | 0.0 (14.03) | -6.0 (15.00) | 2.1 (21.92)
  Week 85: number analyzed (Participants) | 9 | 8 | 5 | 1
  Week 85 | 0.9 (27.78) | -5.2 (7.63) | -3.3 (18.26) | 0.0
  Week 97: number analyzed (Participants) | 4 | 6 | 2 | 0
  Week 97 | -8.3 (6.80) | -2.8 (6.80) | 0.0 (0.00) |
  Week 109: number analyzed (Participants) | 3 | 1 | 2 | 0
  Week 109 | -13.9 (17.35) | 0.0 | 12.5 (5.89) |
  Week 121: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 121 |  | -8.3 |  |
  Week 133: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 133 |  | 0.0 |  |

13. Other Pre Specified Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Breast Cancer Module (QLQ-BR23) at Weeks 5, 9, 17, 25, 33, 41, 49, 61, 73, 85, 97, 109, 121 and 133
Description: EORTC QLQ-BR23 was disease-specific module for breast cancer developed as supplement for EORTC QLQ-C30 that assessed quality of life of participants with breast cancer.Participants self-rated on frequent symptoms or problems reported by participants with breast cancer,e.g., pain/discomfort, body satisfaction, and self-esteem during past week by choosing 1 of 4 possible responses that recorded level of intensity (not at all, a little, quite a bit, and very much) within each dimension.Raw scores were then transformed to 0-100 scale for analysis and interpretation, where higher scores=more level of intensity, as per EORTC guidelines.Participants also self-rated on sexual health/interest during last 4 weeks using same scale. In this outcome measure body image functioning, sexual functioning, systemic therapy side effects, upset by hair loss parameters were assessed by EORTC QLQ-BR23 questionnaire,total score for each parameter ranged from 0-100,where higher scores=more level of intensity.
Time Frame: Baseline; Weeks 5, 9, 17, 25, 33, 41, 49, 61, 73, 85, 97, 109, 121 and 133
Population: ITT population included all the participants randomly assigned to double-blind study treatment. Here, "Overall Number of Participants Analyzed" contributed data to table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for the specified rows and value as "0" indicated no participants filled the questionnaire for the specified reporting group at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 63 | 60 | 60
units on a scale
  Body Image Functioning: Week 5: number analyzed (Participants) | 55 | 57 | 52 | 54
  Body Image Functioning: Week 5 | 1.8 (16.01) | 1.9 (19.10) | -6.1 (13.92) | 2.2 (15.74)
  Body Image Functioning: Week 9: number analyzed (Participants) | 53 | 50 | 40 | 44
  Body Image Functioning: Week 9 | -3.5 (12.91) | -0.2 (17.91) | -3.7 (12.51) | 2.1 (15.58)
  Body Image Functioning: Week 17: number analyzed (Participants) | 43 | 38 | 24 | 31
  Body Image Functioning: Week 17 | -2.9 (20.16) | -3.5 (19.24) | -9.0 (19.34) | 1.3 (13.98)
  Body Image Functioning: Week 25: number analyzed (Participants) | 36 | 33 | 15 | 21
  Body Image Functioning: Week 25 | 2.8 (16.55) | -7.4 (24.24) | -9.4 (16.33) | -0.8 (7.86)
  Body Image Functioning: Week 33: number analyzed (Participants) | 34 | 29 | 9 | 14
  Body Image Functioning: Week 33 | -2.9 (22.08) | -5.7 (17.55) | -1.9 (9.11) | -1.8 (8.12)
  Body Image Functioning: Week 41: number analyzed (Participants) | 29 | 22 | 9 | 12
  Body Image Functioning: Week 41 | -2.5 (18.76) | -1.3 (13.36) | 0.0 (4.17) | 4.2 (14.43)
  Body Image Functioning: Week 49: number analyzed (Participants) | 27 | 21 | 7 | 8
  Body Image Functioning: Week 49 | -2.4 (19.79) | -5.2 (17.57) | -1.2 (3.15) | 1.0 (8.26)
  Body Image Functioning: Week 61: number analyzed (Participants) | 20 | 19 | 7 | 4
  Body Image Functioning: Week 61 | 3.3 (19.94) | -5.7 (15.23) | -4.8 (6.56) | 0.0 (13.61)
  Body Image Functioning: Week 73: number analyzed (Participants) | 14 | 13 | 7 | 4
  Body Image Functioning: Week 73 | -3.2 (29.70) | -3.2 (12.05) | 1.2 (5.75) | 4.2 (10.76)
  Body Image Functioning: Week 85: number analyzed (Participants) | 10 | 8 | 5 | 1
  Body Image Functioning: Week 85 | 8.3 (28.05) | -13.5 (24.78) | 1.7 (3.73) | -16.7
  Body Image Functioning: Week 97: number analyzed (Participants) | 3 | 6 | 2 | 0
  Body Image Functioning: Week 97 | -5.6 (17.35) | -1.4 (3.40) | -4.2 (5.89) |
  Body Image Functioning: Week 109: number analyzed (Participants) | 4 | 1 | 2 | 0
  Body Image Functioning: Week 109 | 0.0 (35.36) | 0.0 | -8.3 (11.79) |
  Body Image Functioning: Week 121: number analyzed (Participants) | 0 | 1 | 0 | 0
  Body Image Functioning: Week 121 |  | 0.0 |  |
  Body Image Functioning: Week 133: number analyzed (Participants) | 0 | 1 | 0 | 0
  Body Image Functioning: Week 133 |  | 0.0 |  |
  Sexual Functioning: Week 5: number analyzed (Participants) | 53 | 52 | 50 | 53
  Sexual Functioning: Week 5 | 1.9 (12.08) | -0.3 (13.40) | 0.3 (17.00) | 1.9 (10.16)
  Sexual Functioning: Week 9: number analyzed (Participants) | 50 | 48 | 38 | 41
  Sexual Functioning: Week 9 | 2.3 (16.15) | -1.4 (16.78) | 1.3 (15.68) | 2.8 (11.73)
  Sexual Functioning: Week 17: number analyzed (Participants) | 40 | 35 | 23 | 29
  Sexual Functioning: Week 17 | 3.3 (15.65) | 0.0 (20.21) | 7.2 (23.48) | 0.6 (12.18)
  Sexual Functioning: Week 25: number analyzed (Participants) | 35 | 32 | 15 | 19
  Sexual Functioning: Week 25 | 1.4 (17.33) | 0.5 (19.16) | 0.0 (25.20) | 1.8 (10.96)
  Sexual Functioning: Week 33: number analyzed (Participants) | 33 | 28 | 9 | 12
  Sexual Functioning: Week 33 | 4.0 (20.43) | 3.0 (12.05) | 7.4 (22.22) | 4.2 (12.56)
  Sexual Functioning: Week 41: number analyzed (Participants) | 28 | 21 | 9 | 10
  Sexual Functioning: Week 41 | 2.4 (23.00) | 0.8 (15.34) | 9.3 (22.22) | 1.7 (9.46)
  Sexual Functioning: Week 49: number analyzed (Participants) | 26 | 20 | 7 | 7
  Sexual Functioning: Week 49 | 7.1 (21.69) | 5.8 (11.18) | 9.5 (26.97) | 0.0 (0.0)
  Sexual Functioning: Week 61: number analyzed (Participants) | 18 | 18 | 7 | 4
  Sexual Functioning: Week 61 | 7.4 (21.56) | 1.9 (20.52) | 7.1 (25.20) | 0.0 (13.61)
  Sexual Functioning: Week 73: number analyzed (Participants) | 14 | 12 | 7 | 4
  Sexual Functioning: Week 73 | 8.3 (16.98) | 2.8 (13.91) | 9.5 (31.71) | 4.2 (8.33)
  Sexual Functioning: Week 85: number analyzed (Participants) | 9 | 7 | 5 | 1
  Sexual Functioning: Week 85 | 7.4 (22.22) | 4.8 (15.85) | -6.7 (27.89) | 0.0
  Sexual Functioning: Week 97: number analyzed (Participants) | 3 | 5 | 2 | 0
  Sexual Functioning: Week 97 | -5.6 (25.46) | 6.7 (9.13) | 16.7 (23.57) |
  Sexual Functioning: Week 109: number analyzed (Participants) | 3 | 1 | 2 | 0
  Sexual Functioning: Week 109 | 0.0 (16.67) | 0.0 | 33.3 (0.00) |
  Sexual Functioning: Week 121: number analyzed (Participants) | 0 | 1 | 0 | 0
  Sexual Functioning: Week 121 |  | 0.0 |  |
  Sexual Functioning: Week 133: number analyzed (Participants) | 0 | 1 | 0 | 0
  Sexual Functioning: Week 133 |  | 0.0 |  |
  Systemic Therapy Side Effects Symptoms: Week 5: number analyzed (Participants) | 55 | 57 | 54 | 54
  Systemic Therapy Side Effects Symptoms: Week 5 | 4.5 (10.59) | 3.7 (10.06) | 7.1 (11.49) | 3.3 (10.82)
  Systemic Therapy Side Effects Symptoms: Week 9: number analyzed (Participants) | 53 | 51 | 42 | 45
  Systemic Therapy Side Effects Symptoms: Week 9 | 7.5 (15.24) | 2.7 (10.24) | 6.5 (11.32) | 3.9 (10.77)
  Systemic Therapy Side Effects Symptoms: Week 17: number analyzed (Participants) | 43 | 38 | 25 | 31
  Systemic Therapy Side Effects Symptoms: Week 17 | 7.5 (10.81) | 2.0 (8.79) | 7.6 (16.61) | 6.0 (12.51)
  Systemic Therapy Side Effects Symptoms: Week 25: number analyzed (Participants) | 37 | 34 | 15 | 21
  Systemic Therapy Side Effects Symptoms: Week 25 | 8.3 (13.90) | 2.3 (7.35) | 5.6 (10.86) | 5.7 (16.05)
  Systemic Therapy Side Effects Symptoms: Week 33: number analyzed (Participants) | 35 | 29 | 9 | 14
  Systemic Therapy Side Effects Symptoms: Week 33 | 6.5 (13.54) | -0.2 (9.74) | 8.5 (7.05) | 5.3 (13.10)
  Systemic Therapy Side Effects Symptoms: Week 41: number analyzed (Participants) | 30 | 22 | 9 | 12
  Systemic Therapy Side Effects Symptoms: Week 41 | 8.4 (10.03) | 1.3 (9.20) | 10.6 (4.63) | 2.0 (10.04)
  Systemic Therapy Side Effects Symptoms: Week 49: number analyzed (Participants) | 27 | 21 | 7 | 8
  Systemic Therapy Side Effects Symptoms: Week 49 | 7.8 (10.18) | 2.5 (11.03) | 9.7 (12.78) | 7.7 (9.84)
  Systemic Therapy Side Effects Symptoms: Week 61: number analyzed (Participants) | 20 | 19 | 7 | 4
  Systemic Therapy Side Effects Symptoms: Week 61 | 7.6 (11.07) | 2.5 (10.45) | 14.7 (10.11) | 4.8 (6.73)
  Systemic Therapy Side Effects Symptoms: Week 73: number analyzed (Participants) | 14 | 13 | 7 | 4
  Systemic Therapy Side Effects Symptoms: Week 73 | 4.9 (11.90) | 4.4 (6.29) | 11.6 (10.95) | -1.2 (5.99)
  Systemic Therapy Side Effects Symptoms: Week 85: number analyzed (Participants) | 10 | 8 | 5 | 1
  Systemic Therapy Side Effects Symptoms: Week 85 | 10.7 (12.58) | 2.4 (8.82) | 9.5 (6.73) | 4.8
  Systemic Therapy Side Effects Symptoms: Week 97: number analyzed (Participants) | 3 | 6 | 2 | 0
  Systemic Therapy Side Effects Symptoms: Week 97 | 8.2 (13.52) | 3.2 (10.29) | 7.1 (10.10) |
  Systemic Therapy Side Effects Symptoms: Week 109: number analyzed (Participants) | 4 | 1 | 2 | 0
  Systemic Therapy Side Effects Symptoms: Week 109 | 14.1 (9.71) | 4.8 | 9.5 (6.73) |
  Systemic Therapy Side Effects Symptoms: Week 121: number analyzed (Participants) | 0 | 1 | 0 | 0
  Systemic Therapy Side Effects Symptoms: Week 121 |  | 9.5 |  |
  Systemic Therapy Side Effects Symptoms: Week 133: number analyzed (Participants) | 0 | 1 | 0 | 0
  Systemic Therapy Side Effects Symptoms: Week 133 |  | 4.8 |  |
  Upset by Hair Loss: Week 5: number analyzed (Participants) | 12 | 11 | 18 | 12
  Upset by Hair Loss: Week 5 | -5.6 (19.25) | 18.2 (31.14) | 0.0 (28.01) | 0.0 (24.62)
  Upset by Hair Loss: Week 9: number analyzed (Participants) | 6 | 10 | 15 | 10
  Upset by Hair Loss: Week 9 | 0.0 (36.51) | 23.3 (31.62) | -6.7 (18.69) | 3.3 (24.60)
  Upset by Hair Loss: Week 17: number analyzed (Participants) | 6 | 7 | 9 | 6
  Upset by Hair Loss: Week 17 | 0.0 (21.08) | 9.5 (16.27) | 3.7 (20.03) | 0.0 (36.51)
  Upset by Hair Loss: Week 25: number analyzed (Participants) | 5 | 7 | 5 | 4
  Upset by Hair Loss: Week 25 | -6.7 (14.91) | 28.6 (35.63) | 26.7 (27.89) | -8.3 (16.67)
  Upset by Hair Loss: Week 33: number analyzed (Participants) | 5 | 5 | 5 | 2
  Upset by Hair Loss: Week 33 | 0.0 (23.57) | -6.7 (14.91) | 20.0 (29.81) | 0.0 (0.00)
  Upset by Hair Loss: Week 41: number analyzed (Participants) | 4 | 3 | 5 | 2
  Upset by Hair Loss: Week 41 | -16.7 (33.33) | 0.00 (0.00) | 13.3 (18.26) | 16.7 (23.57)
  Upset by Hair Loss: Week 49: number analyzed (Participants) | 5 | 2 | 3 | 2
  Upset by Hair Loss: Week 49 | 6.7 (36.51) | 0.0 (0.0) | 11.1 (19.25) | 0.0 (0.0)
  Upset by Hair Loss: Week 61: number analyzed (Participants) | 3 | 2 | 4 | 0
  Upset by Hair Loss: Week 61 | 11.1 (19.25) | 16.7 (23.57) | 25.0 (31.91) |
  Upset by Hair Loss: Week 73: number analyzed (Participants) | 2 | 1 | 5 | 0
  Upset by Hair Loss: Week 73 | 0.0 (0.0) | 0.0 | 40.0 (43.46) |
  Upset by Hair Loss: Week 85: number analyzed (Participants) | 1 | 0 | 3 | 0
  Upset by Hair Loss: Week 85 | 33.3 |  | 0.0 (0.0) |
  Upset by Hair Loss: Week 97: number analyzed (Participants) | 0 | 0 | 1 | 0
  Upset by Hair Loss: Week 97 |  |  | 0.0 |
  Upset by Hair Loss: Week 109: number analyzed (Participants) | 0 | 0 | 2 | 0
  Upset by Hair Loss: Week 109 |  |  | 0.0 (0.0) |
  Upset by Hair Loss: Week 121: number analyzed (Participants) | 0 | 0 | 0 | 0
  Upset by Hair Loss: Week 133: number analyzed (Participants) | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: Number of Participants With Positive Androgen Receptor (AR) Expression by Immunohistochemistry (IHC)
Time Frame: Day 1, 29, 57, 113 and 169
Population: Protocol of this study was amended and data for this outcome measure was not analyzed as per planned analysis.
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first (approximately up to 10.13 years)
Population: Safety population included all the participants who received study drug either in double blind or in open label treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 63 | 60 | 60
Participants
  AEs | 59 | 58 | 58 | 53
  SAEs | 14 | 13 | 10 | 8

16. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events of Grade 3 or Higher Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of the AEs was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Only the participants with treatment-emergent AEs of grade 3 (severe) or higher grade were reported in this outcome measure.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 63 | 60 | 60
Participants | 21 | 16 | 22 | 12

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for clinically significant vital sign abnormalities: Systolic blood pressure (SBP): absolute SBP <90 millimeters of mercury (mmHg) and decrease from baseline (DFB) >30 mmHg, absolute SBP>180 mmHg and increase from baseline (IFB) >40 mmHg, final visit or 2 consecutive visits SBP >=20 mmHg change from baseline (CFB), most extreme post-baseline SBP >=140 mmHg, most extreme post-baseline SBP >=180 mmHg, most extreme SBP >=140 mmHg and >=20 mmHg CFB, most extreme SBP >=180 mmHg and >=20 mmHg CFB; diastolic blood pressure (DBP): absolute DBP > 105 mmHg and IFB >30 mmHg, absolute DBP <50 mmHg and DFB >20 mmHg, final visit or 2 consecutive visits DBP >=15 mmHg CFB, most extreme post-baseline DBP >=90 mmHg, most extreme post-baseline DBP >=105 mmHg, most extreme DBP >=90 mmHg and >=15 mmHg CFB, most extreme DBP >=105 mmHg and >=15 mmHg CFB; heart rate <50 beats per minute (BPM) and DFB >20 BPM or heart rate >120 BPM and IFB >30 BPM.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 63 | 60 | 60
Participants
  Blood pressure | 38 | 39 | 43 | 25
  Heart rate | 0 | 2 | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory tests included hematology (hematocrit, hemoglobin, platelet count, red blood cell count, total neutrophils [absolute] and white blood cell count with differential) and serum chemistry (albumin, alkaline phosphatase, alanine aminotransferase [ALT], aspartate transaminase [AST], blood urea nitrogen and creatinine, calcium, sodium, potassium, chloride, glucose (non-fasting), lactate dehydrogenase, magnesium, phosphorus/phosphate, total bilirubin, total bicarbonate, total protein and uric acid). Clinically significant abnormality evaluation was based on clinical investigator's judgment.
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first (up to 3 years)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 63 | 60 | 60
Participants | 0 | 0 | 0 | 0

19. Other Pre Specified Outcome: Progression Free Survival (PFS): By Electronic Data Capture (EDC)
Description: PFS was defined as the time in months from randomization to the first documentation of PD or death on study due to any cause, whichever occurred first. PD according to RECIST 1.1 was defined >=20 % increase in the sum of diameters of the target lesions taking as a reference the smallest sum recorded since the start of treatment or unequivocal progression in non-target lesions or the appearance of 1 or more new lesions. The analysis of PFS was based on investigator assessment of disease progression. Participants who were not known to have had a PFS event at the analysis date were censored at last tumor assessment date prior to data cutoff or date of new treatment initiation, whichever occurred first. Cht 1: Enz + Exe = Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg; Cht 2: Enz + Exe= Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg
Time Frame: as for outcome 1
Population: Analysis was performed on all randomized participants. Randomization to cohort was based on participant's exposure to advance setting hormonal therapy. Initial randomization was done by IWRS. Later, upon detailed data entry in EDC, it was determined 1 participant was incorrectly assigned to Cht1:Enz+Exe by IWRS,hence counted in Cht2:Enz+Exe by EDC.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 62 | 64 | 61 | 60
Months | 11.8 [7.3 to 14.6] | 5.8 [3.5 to 10.9] | 3.6 [1.9 to 5.6] | 3.9 [2.6 to 5.4]
Statistical Analysis 1: Comparison: Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 1: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.7378, Stratified log-rank; Hazard Ratio (HR) = 0.928, 95% CI 2-sided [0.599 to 1.438]
Statistical Analysis 2: Comparison: Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 2: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.8817, Stratified log-rank; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.632 to 1.483]

20. Other Pre Specified Outcome: Progression Free Survival (PFS): Diagnostic Positive (DX+) Population By Electronic Data Capture (EDC)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
Number analyzed (Participants) | 23 | 26 | 16 | 20
Months | 16.9 [11.0 to NA] — Upper limit of 95% confidence interval was not reached due to insufficient number of events at the time of data cutoff (23 Sep 2016). | 4.3 [1.9 to 10.9] | 6.0 [3.5 to 16.6] | 5.3 [1.8 to 6.7]
Statistical Analysis 1: Comparison: Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 1: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.1270, Stratified log-rank; Hazard Ratio (HR) = 0.522, 95% CI 2-sided [0.224 to 1.217]
Statistical Analysis 2: Comparison: Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg vs Cohort 2: Placebo + Exemestane 25 mg; Hazard ratio was based on stratified Cox regression model; Test type: Other; p = 0.0359, Stratified log-rank; Hazard Ratio (HR) = 0.370, 95% CI 2-sided [0.143 to 0.961]

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first (up to 10.13 years)
Description: Same event may appear as both an adverse event (AE) and a serious AE, but they are distinct events. Event may be categorized as serious in one participant and as non-serious in another, or one may have experienced both serious and non-serious event during study. AEs and all-cause mortality were collected and evaluated for safety population.
Arm/Group | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 1: Placebo + Exemestane 25 mg | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg | Cohort 2: Placebo + Exemestane 25 mg
All-Cause Mortality (participants affected / at risk) | 2/62 | 8/63 | 3/60 | 2/60
Serious Adverse Events (participants affected / at risk) | 14/62 | 13/63 | 10/60 | 8/60
Other Adverse Events (participants affected / at risk) | 59/62 | 57/63 | 57/60 | 52/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg (N=62) | Cohort 1: Placebo + Exemestane 25 mg (N=63) | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg (N=60) | Cohort 2: Placebo + Exemestane 25 mg (N=60)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 0 | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0 | 0
CHILLS (General disorders) | 1 | 0 | 0 | 0
DISEASE PROGRESSION (General disorders) | 0 | 1 | 1 | 0
FACIAL PAIN (General disorders) | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 0 | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0 | 0
PAIN (General disorders) | 1 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 0 | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 0
BREAST CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 0
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OPTIC NERVE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
MASTICATION DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
CONTRALATERAL BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BRACHIAL PLEXOPATHY (Nervous system disorders) | 0 | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 1 | 0 | 0
EMBOLIC STROKE (Nervous system disorders) | 0 | 0 | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1 | 0 | 0
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 0 | 0 | 0 | 1
SPEECH DISORDER (Nervous system disorders) | 0 | 0 | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 1 | 0 | 0
STATUS EPILEPTICUS (Nervous system disorders) | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 0
DELIRIUM (Psychiatric disorders) | 0 | 0 | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Enzalutamide 160 mg + Exemestane 50 mg (N=62) | Cohort 1: Placebo + Exemestane 25 mg (N=63) | Cohort 2: Enzalutamide 160 mg + Exemestane 50 mg (N=60) | Cohort 2: Placebo + Exemestane 25 mg (N=60)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 1 | 6 | 3
CONSTIPATION (Gastrointestinal disorders) | 11 | 7 | 8 | 8
DIARRHOEA (Gastrointestinal disorders) | 14 | 10 | 7 | 11
DYSPEPSIA (Gastrointestinal disorders) | 1 | 6 | 5 | 4
NAUSEA (Gastrointestinal disorders) | 24 | 10 | 18 | 11
VOMITING (Gastrointestinal disorders) | 11 | 7 | 6 | 3
ASTHENIA (General disorders) | 9 | 7 | 6 | 4
FATIGUE (General disorders) | 24 | 23 | 21 | 13
URINARY TRACT INFECTION (Infections and infestations) | 2 | 3 | 1 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 | 2 | 4
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 4 | 2 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 6 | 6 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 11 | 10 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 | 6 | 4 | 11
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 7 | 4 | 3 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 8 | 3 | 5
DIZZINESS (Nervous system disorders) | 7 | 4 | 5 | 2
HEADACHE (Nervous system disorders) | 9 | 6 | 9 | 10
ANXIETY (Psychiatric disorders) | 6 | 4 | 2 | 1
INSOMNIA (Psychiatric disorders) | 5 | 4 | 5 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 2 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 5 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 8 | 4 | 5 | 2
HOT FLUSH (Vascular disorders) | 19 | 14 | 14 | 9
HYPERTENSION (Vascular disorders) | 8 | 3 | 2 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 1 | 1 | 3
INFLUENZA (Infections and infestations) | 3 | 4 | 1 | 2
PARAESTHESIA (Nervous system disorders) | 4 | 2 | 2 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 4 | 3 | 0 | 1
AMNESIA (Nervous system disorders) | 4 | 0 | 1 | 1
DEPRESSED MOOD (Psychiatric disorders) | 1 | 0 | 4 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 2 | 4 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.